CLINICAL TRIAL: NCT03762031
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Dose Escalation Study Designed to Evaluate the Safety and Pharmacokinetics of Intravenously Administered Superoxide Dismutase Mimetic GC4711 in Healthy Volunteers
Brief Title: A Study Designed to Evaluate the Safety and Pharmacokinetics of Intravenously Administered Superoxide Dismutase Mimetic GC4711 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTI-4711-002
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- GC4711 30mg (Experimental)
  Interventions: Drug: GC4711 30mg
- GC4711 60mg (Experimental)
  Interventions: Drug: GC4711 60mg
- GC4711 90mg (Experimental)
  Interventions: Drug: GC4711 90mg
- GC4711 120mg (Experimental)
  Interventions: Drug: GC4711 120mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- GC4711 75mg (Experimental)
  Interventions: Drug: GC4711 75mg
- GC4711 105mg (Experimental)
  Interventions: Drug: GC4711 105mg

INTERVENTIONS:
Drug: GC4711 30mg — single dose given via a 15 minute intravenous infusion
  Arms: GC4711 30mg
Drug: GC4711 60mg — single dose given via a 15 minute intravenous infusion
  Arms: GC4711 60mg
Drug: GC4711 90mg — single dose given via a 15 minute intravenous infusion
  Arms: GC4711 90mg
Drug: GC4711 120mg — single dose given via a 15 minute intravenous infusion
  Arms: GC4711 120mg
Drug: Placebo — single dose of normal saline given via a 15 minute intravenous infusion
  Arms: Placebo
Drug: GC4711 75mg — single dose given via a 15 minute intravenous infusion
  Arms: GC4711 75mg
Drug: GC4711 105mg — single dose given via a 15 minute intravenous infusion
  Arms: GC4711 105mg

SUMMARY:
The study will be a Phase 1, randomized, double-blind, placebo-controlled, single dose escalation study designed to evaluate the safety and PK of intravenously administered superoxide dismutase mimetic GC4711 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women between 18 and 50 years
2. Subjects who provide written informed consent
3. Body Mass Index (BMI) of 18 to 32 kg/m2 and weighing at least 50 kg
4. Subjects in general good health
5. Blood pressure and pulse within normal limits
6. Male subjects must practice effective contraception
7. Female subjects must:

   * Have a negative serum pregnancy test during
   * Be non-lactating;
   * Be at least 2 years postmenopausal, surgically sterile, or practicing effective contraception.

Exclusion Criteria:

1. History of clinically significant illness or medical history which would preclude them from the study.
2. Known contraindication, hypersensitivity and/or allergy to study drugs
3. Use of any prescription or over-the-counter medication within one week prior to study drug administration
4. Anticipated need for any medication during the study
5. Use of nitrates or erectile dysfunction drugs such as phosphodiesterase type 5 (PDE 5) inhibitors
6. Use of other drugs that may, in the judgment of the Investigator, create a risk for a precipitous decrease in blood pressure
7. Presence of orthostatic hypotension at screening
8. Use of any vitamin or mineral supplement 24 hours before dosing or throughout study
9. Positive human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C (HCV)
10. Known history of substance abuse, drug addiction, or alcoholism within 3 years
11. Anticipated inability to abstain from alcohol, tobacco, or caffeine use from 48 hours before the administration of study drug and throughout the the study;
12. Positive drug and alcohol toxicology screens during Screening
13. History of smoking or any use of a tobacco product within 6 months
14. Donation of blood or blood products within 30 days before Baseline and throughout the study;
15. Mentally unstable or incapable of being compliant with the protocol
16. Receipt of an investigational test substance within 3 months before the administration of study drugs, or anticipated receiving any study drugs
17. Subject has previously participated in this study, or in a prior Galera study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events and Laboratory Abnormalities | From randomization through study completion (estimated up to 3 days)
  Number of Participants With Treatment-Emergent Adverse Events and/or Laboratory Abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Jon Holmlund, MD, Study Chair — Galera Therapeutics, Inc.
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No